CLINICAL TRIAL: NCT04586283
Title: Does Maternal Prone Position Affect Maternal Cardiorespiratory Status or the Fetal Heart Rate?
Brief Title: Does Prone Position Alter Maternal Cardiorespiratory Status?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Dr Alexander Heazell, Professor of Obstetrics, University of Manchester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRAS240071
Record Dates: First submitted 2020-09-22; First posted 2020-10-14 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Pregnancy-Related Condition, Unspecified
Keywords: Maternal prone position; Cardiac output; Fetal heart rate; Cardiotocography; Maternal anxiety

STUDY DESIGN:
Intervention Model Description: Cohort study
Masking Description: As the study involves examination of cardiorespiratory indices in different maternal positions investigators cannot be blind to the participants' position.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Maternal Prone Position (Experimental): Participants will initially be assessed in left-lateral position for 20 minutes. Participants will then be asked to lie in a prone position for 30 minutes supported by a specially designed pillow. Participants will then return to a left-lateral position for 20 minutes.
  Interventions: Other: Maternal prone position

INTERVENTIONS:
Other: Maternal prone position — Women will be asked to lie in a prone position supported by a specially designed cushion for 30 minutes.

SUMMARY:
During pregnancy women may need or choose to undergo physical therapies such as physiotherapy, massage or osteopathy. Recent findings from studies of mothers who had a stillbirth in late pregnancy found that the position in which women went to sleep in was linked to stillbirth, as was the frequency of day time naps. This link is thought to be due to changes in mother's blood flow from her heart when lying flat leading to changes in the amount of oxygen going to her baby. This raise concerns that spending extended periods laid flat could be detrimental to baby's health. However, it is not known whether lying flat for extended periods for physical therapies could also alter a baby's heart rate or levels of oxygen. One small study of 33 women from Brazil found that there were no differences in a mother's heart rate, blood pressure, oxygen saturation or baby's heart rate. But there were changes in mother's breathing rate and systolic blood pressure when a mother laid on her front. All the women reported feeling comfortable lying flat (on a bent surface). However, in this study women only spent 6 minutes in each position which is less than a woman would be expected to spend lying in a position for a session of physical therapy. The investigators plan a study to assess whether using a device to support a prone position (Anna cushion) would be associated with changes in mother's heart rate, blood pressure, breathing rate and blood oxygen levels and baby's heart rate. The investigators will also ask about mother's levels of comfort while she is laid in the prone position. The findings of this study will give an indication whether supporting a mother to lie in a prone position for physical therapies is safe and comfortable.

DETAILED DESCRIPTION:
Women frequently experience lower-back or pelvic pain during pregnancy. This may lead to a need for physical therapies such as physiotherapy, osteopathy or massage in late pregnancy. Several case-control studies, and a recent individual patient data meta-analysis has demonstrated an association between going to sleep position and late stillbirth (a greater than 2-fold increased risk with going to sleep supine) and increased frequency of daytime naps. This is thought to be related to maternal haemodynamic changes when a mother lies supine in late pregnancy which decreases cardiac output and uterine blood flow. These changes are accompanied by alterations in fetal behaviour which are consistent with a reduction in oxygenation. This observation raises concerns that spending extended periods laid flat could be detrimental to baby's health. However, it is not known whether lying flat for extended periods for physical therapies could also alter a baby's heart rate or levels of oxygen. One small study of 33 women from Brazil which randomised the order of maternal positions found that there were no differences in a mother's heart rate, blood pressure, oxygen saturation or baby's heart rate between a supine, lateral and prone position (bent over a concave couch). However, there were observed changes in mother's breathing rate and systolic blood pressure when a mother laid on her front. Nevertheless, all the women reported feeling comfortable lying flat (on a bent surface). However, in this study women only spent 6 minutes in each position which is less than a woman would be expected to spend lying in a position for a session of physical therapy. Therefore, further work is required to determine whether spending extended periods laid prone is safe for mother and baby.

The co-investigator (Karli Büchling) has developed a cushion to support mothers in a prone position (Anna cushion). This study will investigate whether adopting this position supported by the cushion is associated with changes in mother's heart rate, blood pressure, breathing rate and blood oxygen levels and fetal heart rate as assessed by the cardiotocograph. The investigators will also ask about mother's levels of comfort while she is laid flat. The findings of this study will give an indication whether supporting a mother to lie in a prone position for physical therapies is safe and comfortable.

ELIGIBILITY:
Inclusion Criteria:

* Viable singleton pregnancy ≥28 weeks' gestation
* No fetal anomalies according to Fetal Anomaly Screening Programme definition
* Ability to give written informed consent
* Maternal Age >16 years

Exclusion Criteria:

* Unable to read English (as the survey instruments are only available in English)
* Multiple pregnancy
* Pre-existing maternal cardiovascular or respiratory disease
* Fetal anomaly
* Contraindication to lying prone (severe pain etc.)
* Allergy to self-adhesive electrodes used for standard electrocardiography (ECG)
* Unable to give written informed consent

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnant women
Enrollment: 21 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-05-16 (Actual)

PRIMARY OUTCOMES:
Maternal cardiac output at Baseline | At baseline
  Maternal cardiac output as assessed by non-invasive cardiac monitoring.
Change in maternal cardiac output | After 30 minutes in prone position
  Maternal cardiac output as assessed by non-invasive cardiac monitoring in prone position. Change calculated as Maternal cardiac output after 30 minutes in prone position - baseline cardiac output.

SECONDARY OUTCOMES:
Maternal heart rate at baseline | At baseline
  Maternal heart rate as assessed by non-invasive monitoring (as beats per minute).
Change in maternal heart rate | After 30 minutes in prone position
  Maternal heart rate as assessed by non-invasive monitoring (as beats per minute) in prone position. Change calculated as Maternal heart rate after 30 minutes in prone position - baseline heart rate.
Maternal respiratory rate | At baseline
  Maternal respiratory rate as assessed by counting respirations (per minute)
Change in maternal respiratory rate | After 30 minutes in prone position
  Maternal respiratory rate as assessed by counting respirations (per minute) in prone position. Change calculated as Maternal respiratory rate after 30 minutes in prone position - baseline respiratory rate.
Maternal blood pressure | At baseline
  Both maternal systolic and diastolic blood pressure as assessed noninvasive blood pressure monitoring
Change in maternal blood pressure | After 30 minutes in prone position
  Both maternal systolic and diastolic blood pressure as assessed noninvasive blood pressure monitoring in prone position. Change calculated as maternal systolic blood pressure after 30 minutes in prone position - baseline systolic blood pressure or maternal diastolic blood pressure after 30 minutes in prone position - baseline diastolic blood pressure.
Oxygen saturation | At baseline
  Oxygen saturation measured by pulse oximetry
Change in oxygen saturation | After 30 minutes in prone position
  Oxygen saturation measured by pulse oximetry in prone position. Change calculated as Maternal oxygen saturation after 30 minutes in prone position - baseline oxygen saturation.
Fetal heart rate | Baseline
  Fetal wellbeing assessed by continuous cardiotocography which will report baseline heart rate, variability, the presence of accelerations or decelerations.
Change in fetal heart rate | Afer 30 minutes in prone position
  Fetal wellbeing assessed by continuous cardiotocography which will report baseline heart rate, variability, the presence of accelerations or decelerations.

OTHER OUTCOMES:
Maternal Anxiety | Before the experimental protocol
  Maternal anxiety will be assessed using the State Trait Anxiety Index (scores range from 20-80, where higher scores indicate greater anxiety).
Maternal Anxiety | Immediately after the completion of the experimental protocol
  Maternal anxiety will be assessed using the State Trait Anxiety Index (scores range from 20-80, where higher scores indicate greater anxiety).
Maternal comfort as assessed by visual analogue scale | Before the experimental protocol
  Maternal comfort as assesed by a visual analogue scale from 0-10. Higher scores indicate greater discomfort.
Maternal comfort as assessed by visual analogue scale | Immediately after the completion of the experimental protocol
  Maternal comfort as assesed by a visual analogue scale from 0-10. Higher scores indicate greater discomfort.
Maternal comfort as assessed by self-reported questionnaire | Immediately after the completion of the experimental protocol
  Maternal comfort as assessed by self-reported questionnaire using Likert scales (from 1-5, where higher scores indicate greater agreement with the statement) and free-text responses

CONTACTS AND LOCATIONS:
Locations (1):
- Manchester University NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There is currently no plans to make individual participant data available to other researchers.

REFERENCES:
- [Derived] Ormesher L, Catchpole J, Peacock L, Pitt H, Fabian-Hunt A, Hayes D, Popp C, Carson JM, van Loon R, Warrander L, Buchling K, Heazell AEP. The effect of prone positioning on maternal haemodynamics and fetal wellbeing in the third trimester-A primary cohort study with a scoping review. PLoS One. 2023 Oct 11;18(10):e0287804. doi: 10.1371/journal.pone.0287804. eCollection 2023. PMID 37819872